CLINICAL TRIAL: NCT01991145
Title: Safety and Efficacy of Allogeneic Umbilical Cord Blood Therapy Combined With Erythropoietin in Children With Cerebral Palsy: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Allogeneic UCB Therapy With EPO in Children With CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, MD, PhD (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); LG Life Sciences (Industry); Chong Kun Dang Pharmaceutical (Industry); CHA University (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, MD, PhD, Professor of CHA University, M.D., Ph.D., Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCBnEPOinCP
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Umbilical Cord Blood; Erythropoietin; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- UCB and EPO (Experimental): UCB + EPO + Rehabilitation
  Interventions: Procedure: Umbilical Cord Blood therapy; Biological: Erythropoietin alfa; Other: Rehabilitation
- UCB and placebo EPO (Active Comparator): UCB + placebo EPO + Rehabilitation
  Interventions: Procedure: Umbilical Cord Blood therapy; Other: Rehabilitation; Biological: Placebo EPO
- placebo UCB and EPO (Active Comparator): placebo UCB + EPO + Rehabilitation
  Interventions: Biological: Erythropoietin alfa; Other: Rehabilitation; Procedure: Placebo UCB
- placebo UCB and placebo EPO (Placebo Comparator): placebo UCB + placebo EPO + Rehabilitation
  Interventions: Other: Rehabilitation; Procedure: Placebo UCB; Biological: Placebo EPO

INTERVENTIONS:
Procedure: Umbilical Cord Blood therapy — HLA (Human Leukocyte Antigen) typing
  Arms: UCB and EPO; UCB and placebo EPO
Biological: Erythropoietin alfa
  Other Names: Espogen (LG Life Science Ltd.)
  Arms: UCB and EPO; placebo UCB and EPO
Other: Rehabilitation — Active rehabilitation
Procedure: Placebo UCB
  Arms: placebo UCB and EPO; placebo UCB and placebo EPO
Biological: Placebo EPO
  Arms: UCB and placebo EPO; placebo UCB and placebo EPO

SUMMARY:
This randomized controlled study aims to evaluate the efficacy and safety of allogeneic umbilical cord blood therapy combined with erythropoietin for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a group of neurodevelopmental conditions with abnormal movement and posture resulted from a non-progressive cerebral disturbance. It is the most common cause of motor disability in childhood. Most therapies are palliative rather than restorative. Umbilical cord blood (UCB) and erythropoetin (EPO) may be used as restorative approach for children with CP.

Many experimental animal studies have revealed that UCB is beneficial to improve and repair neurological injuries. EPO is also known to have neuroprotective effects.

Based on animal studies and some clinical trials, UCB is suggested as a potential therapy for children with CP. EPO is combined to add synergistic effects to UCB therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy
* Age of ≥10 months and ≤6 years
* Mismatch in HLA-A, B, and DR ≤2, and total nucleated cell count ≥3x107/kg. If the cell count is less than given values, more than 1 unit could be used.
* Hemoglobin ≤13.6 g/dL
* Decision of participation in the study by and acquisition of informed consent from the subject's representative
* Willingness and ability to be hospitalized according to the schedule specified in the protocol and continue the study for 12 months after study entry

Exclusion Criteria:

* Current aspiration pneumonia
* Known genetic disease
* History of hypersensitivity reaction to any study drugs pertinent to the study
* History of participation in any other study with stem cell
* Prior treatment with EPO within 3 months prior to study entry
* Known coagulopathy with family history of thrombosis or medical history of recurrent thrombosis
* Patient with severe seizure disease who has clinical convulsion despite combination therapy with 3 or more agents
* Uncontrolled hypertension defined as systolic blood pressure >115 mmHg and/or diastolic blood pressure >70 mmHg
* Hepatic impairment defined as asparate aminotransferase (AST) >55 IU/L and/or alanine aminotransferase (ALT) >45 IU/L
* Renal impairment defined as creatinine (Cr) ≥1.2 mg/dL
* Absolute neutrophil count ≤500/dL
* Presence of diagnosed or suspected malignant tumor and/or hematologic malignancy
* Non-compliance with study visits specified in the protocol or unwillingness of care-giver due to lack of understanding of the patient

Ages: 10 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2017-06-24 (Actual); Study Completion 2017-06-24 (Actual)

PRIMARY OUTCOMES:
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months - 6 months - 12months
  GMFM (Gross Motor Function Measure) is a standardized measurement tool for assessing gross motor function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100, higher value means better gross motor function).
Changes in Motor Performance | Baseline - 1 month - 3 months - 6 months - 12 months
  GMPM (Gross Motor Performance Measure) is a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, higher value means better motor quality).
Changes in Cognitive Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Mental Scale (range: 0~178; worst: 0, best: 178)
Changes in Motor Neurodevelopmental Outcome | Baseline - 1 month - 3 months - 6 months - 12 months
  Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor Scale (range: 0~112; worst: 0, best: 112)

SECONDARY OUTCOMES:
Changes in Gross Motor Function Classification System | Baseline - 1 month - 3 months - 6 months - 12 months
  GMFCS (Gross Motor Function Classification System) is a five-level classification system based on self-initiated movement, with emphasis on sitting, transfers, and mobility (level I: walks without limitations, ll: walks with limitations, III: walks using a hand-held mobility device, IV: self-mobility with limitations, V: transported in a manual wheelchair).
Changes in Functional Independence in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher score means more independent performance in daily activities.
Changes in Functional Performance in Daily Activities | Baseline - 1 month - 3 months - 6 months - 12 months
  Pediatric Evaluation of Disability Inventory (PEDI) is used to assess functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best). PEDI consists of 2 scales such as Functional Skill Scale (FSS) and a Caregiver Assistance Scale (CAS) and each scale is composed of 3 domains including self care, mobility, and social function.
Changes in Upper Extremity Function | Baseline - 1 month - 3 months - 6 months - 12 months
  QUEST (Quality of Upper Extremity Skills Test) is a standardized measurement tool for assessing upper extremity function consisting of sub-scales; dissociated movement, grasps, weight bearing, and protective extension. QUEST ranges from 0 (or below 0 in grasp section) to 100 and higher values mean better upper extremity function.
Changes in Visual Perception Test | Baseline - 1 month - 3 months - 6 months - 12 months
  Visual perception function will be assessed with one of 3 tools such as DTVP (Developmental Test of Visual Perception), MVPT (Motor-free Visual Perception Test), and VMI (Visual-Motor Integration, Visual Perception and Motor Coordination). Higher value means better visual perception ability.
Changes in Selective Movement of Lower Extremity | Baseline - 1 month - 3 months - 6 months - 12 months
  SCALE (Selective Control Assessment of Lower Extremity) is a measurement tool of selective movement of hip, knee, ankle, subtalar joint and toes. Selective voluntary motor control is graded at each joint as normal (2 points), impaired (1 point) or unable (0 point).
Changes in Spasticity | Baseline - 1 month - 3 months - 6 months - 12 months
  Muscle spasticity of biceps, hip adductors, hamstrings and heel cords is graded according to modified Ashworth scale (MAS).
Changes in Dynamic Component of Spasticity | Baseline - 1 month - 3 months - 6 months - 12 months
  Dynamic component of spasticity in bilateral hamstrings is graded using modified Tardieu scale (MTS).
Changes in Muscle Strength | Baseline - 1 month - 3 months - 6 months - 12 months
  Muscle strength is measured using summated scores of manual muscle test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160). Higher score means stronger muscle power.
Changes in Brain MRI | Baseline - 12 months
  Diffusion Tensor Image (DTI) of brain MRI (magnetic resonance imaging) provides quantitative information about the microscopic integrity of white matter. White matter normally possesses a high degree of diffusion anisotropy than gray matter. Fractional anisotropy (FA) will be measured and it ranges from 0 to 1. Higher FA value means more integrity of white matter.
Changes in Brain 18F-FDG PET | Baseline - 12 months
  18F-FDG PET (Positron emission tomography with fluorine-18-fluorodeoxyglucose) imaging will be performed twice prior to and 12 months after UCB therapy.
Changes in EEG | Baseline - 12 months
  Electroencephalography (EEG) will be performed twice prior to and 12 months after UCB therapy.
Changes in EP | Baseline - 12 months
  Median, tibial somatosensory evoked potential (SEP), visual evoked potential (VEP), auditory evoked potential (AEP) will be performed twice prior to and 12 months after UCB therapy.
Number of adverse events and participants with those adverse events | 12 months
  The numbers of adverse events and subjects with those serious adverse events within each group; A serious adverse event is any untoward medical occurrence that at any dose: results in death or is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or causes a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: MinYoung Kim, M.D., Ph.D., Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Min K, Suh MR, Cho KH, Park W, Kang MS, Jang SJ, Kim SH, Rhie S, Choi JI, Kim HJ, Cha KY, Kim M. Potentiation of cord blood cell therapy with erythropoietin for children with CP: a 2 x 2 factorial randomized placebo-controlled trial. Stem Cell Res Ther. 2020 Nov 27;11(1):509. doi: 10.1186/s13287-020-02020-y. PMID 33246489